CLINICAL TRIAL: NCT05824208
Title: PRENAYOGA: Exploratory Feasibility Study of Bi-weekly Pregnancy Yoga-based Sessions for Ethnic Minority Women
Acronym: PRENAYOGA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HR/DP-22/23-34528
Record Dates: First submitted 2023-03-24; First posted 2023-04-21 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-03

CONDITIONS: Prenatal Stress; Pregnancy Related; Complementary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bi-weekly pregnancy yoga-based sessions for 8 weeks (Experimental)
  Interventions: Behavioral: PRENAYOGA - prenatal yoga

INTERVENTIONS:
Behavioral: PRENAYOGA - prenatal yoga — The intervention is a prenatal yoga module developed for prenatal women. Intervention details: bi-weekly yoga classes (60 minutes of duration) will be delivered in person in a yoga studio in London for 8 consecutive weeks. Participants will be provided with yoga mats, blocks, bolsters and yoga straps at the studio. The class will be adapted to pregnancy and for all levels of ability, focusing on slow movements and body awareness. The content of the class will include loosening exercises (warm up exercises), simple postures (standing, balancing, sitting, kneeling, supine and restorative poses), breathing exercises and meditation. Classes will be delivered by an internationally certified and trained yoga teacher and will be accompanied by soft instrumental music.

SUMMARY:
Depression and anxiety are the most prevalent psychiatric disorders in the perinatal period. A recent report found that nearly 50% of new mothers in London (where 40% of the population is of ethnic minority background) display symptoms of postnatal depression (PND).

A 2022 report by the London School of Economics (LSE) found that treating maternal mental illness could save the National Health Service (NHS) £52 million over 10 years; in 2014, the LSE calculated that two-thirds of that cost is linked to adverse child development.

Prenatal depression results in adverse outcomes for the mother and infant, which are also linked to the impact of postnatal depression on the emotional relationship and attachment between the mother and the child. The major risk for developing depression postnatally is a history of depression, either in the lifetime or during pregnancy.

Several studies highlight that antenatal depression rates are higher in ethnic minority women. However, the percentage of ethnically diverse women in most studies on perinatal depression is negligible. Additionally, ethnic minority women are less represented in perinatal mental health therapeutic settings.

Preliminary evidence indicates prenatal yoga reduces anxiety and depression and improves mother-foetal attachment. Ethnic minorities support mind-body interventions such as yoga and may be more likely to engage in community-based activities than traditional antenatal classes.

An 8-week feasibility study will assess the feasibility and acceptability of a yoga-based intervention for ethnic minority women in London.

DETAILED DESCRIPTION:
This exploratory feasibility study intends to understand participants' experiences and implementation considerations of an evidence-based, stakeholder-co-designed prenatal yoga intervention.

Participants will be recruited through signposting in the community and social media. Potential participants will complete an online form store on the study-specific SharePoint where they will include their name, date of birth, due date, mobile number, e-mail address, home address, GP/midwife contact details, frequency of previous yoga practice and availability for the study. This information will allow researchers to assess for eligibility and gather contact details for baseline assessment. The ICF and PIS will be sent to participants who fulfil the eligibility criteria. If participants do not enrol on the study, their information will be deleted.

Once they agree to be part of the study and basic demographics are collected on Zoom, participants will be sent, via e-mail, questionnaires to complete (on their phones or laptops) to evaluate their mental health, social support and attachment to the baby. These questionnaires are surveys that can be answered quickly and allow researchers to quantify changes in psychological states over time. Implementation questionnaires to understand how the intervention can be tested in future large-scale studies will also be collected on REDCap. Attendance and enrolment rates will also be collected for adherence and uptake implementation measures.

Questionnaires will be again completed at week 4 (midpoint of the study), week 8 (end of study), at 8 weeks postpartum and 6 months postpartum. There will be a 2-week leeway for questionnaire completion by participants.

Salivary cortisol samples will be collected at the beginning and end of sessions 1 and 8 to assess in-person changes in cortisol outputs during the yoga sessions.

Changes in participants' depression, anxiety, social support, maternal-foetal attachment and cortisol levels will be quantified to understand if the yoga programme may impact these aspects.

Participants will be asked to provide qualitative data on their views of the intervention and the study in the following formats:

* Focus group in the last week of the study on the experience of the intervention and barriers/facilitators
* Interviews with participants who attend less than 50% of sessions or withdraw from the study on their experience of the intervention and barriers/facilitators of the intervention.

Interviews and focus groups are optional (this is mentioned in the PIS and ICF).

Questions for focus groups and interviews will be around the overall experience of the intervention, expectations, acceptability, reasons for missed sessions, adoption, preference for sessions in person/online, willingness to undergo randomisation on an RCT, and acceptability of the questionnaires and samples. In the focus groups, I will also ask about facilitators and barriers, the appropriateness of the sessions, how feasible it was for them to attend the sessions and any factors that may affect the long-term scalability/sustainability of the yoga sessions.

Intervention: bi-weekly yoga classes (60 minutes duration, twice per week) will be delivered in person in a yoga studio in London for 8 consecutive weeks. Participants will be provided with yoga mats, blocks, bolsters and yoga straps at the studio. The class will be adapted to pregnancy and for all levels of ability, focusing on slow movements and body awareness. The content of the class will include loosening exercises (warm-up exercises), simple postures (standing, balancing, sitting, kneeling, supine and restorative poses), breathing exercises and meditation. Classes will be delivered by an internationally certified and trained yoga teacher and will be accompanied by soft instrumental music.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age: week 20 of gestation or over, at the first session.
* Over 18 years of age.
* Basic understanding of English.
* Able to travel to the sessions.
* Belonging to an ethnic minority group (self-identified) other than White.

Exclusion Criteria:

- Physical or mental health diagnosis that would prevent them from attending yoga sessions, as per their healthcare professional's advice (self-reported).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-03-28 (Actual); Primary Completion 2023-06-03 (Actual); Study Completion 2023-06-17 (Actual)

PRIMARY OUTCOMES:
To assess the acceptability of the intervention | End of intervention (week 8).
  Total score of the Acceptability of Intervention Measure (AIM). The Acceptability of Intervention Measure (AIM) has a scale range of 1-5, with higher scores indicating greater acceptability.

SECONDARY OUTCOMES:
To assess reasons for perceived acceptability of the intervention | End of intervention (week 8).
  Focus groups
To assess uptake/reach of the intervention | End of intervention (week 8).
  Number of eligible women that sign up to the intervention
To assess the appropriateness of the intervention | End of intervention (week 8).
  Total score of the Intervention Appropriateness Measure (IAM). The Intervention Appropriateness Measure (IAM) has a scale range of 1-5, with higher scores indicating greater appropriateness of the intervention.
To assess the feasibility of the intervention | End of intervention (week 8).
  Total score of the Feasibility of Intervention Measure (FIM). FIM has a scale range of 1-5, higher scores indicate greater feasibility of the intervention, assessing the practicality and potential for success of an intervention in a particular setting or population based on factors such as ease of implementation, cost-effectiveness, and stakeholder acceptability.
To assess intervention adherence and attrition rates | End of intervention (week 8).
  Data on the overall adherence to the intervention, number of drops-outs each week.
To assess the effects of quality of life | Start (baseline) and end of intervention (week 8).
  EQ5D-5L (quality of life measure). The EQ5D-5L is a quality of life measure that can be presented as EQ VAS and EQ-5D-5L index value.
To assess factors affecting the sustainability and scalability of the intervention | End of intervention (week 8).
  Focus groups
To assess the effectiveness of group prenatal yoga to increase mother-foetal attachment | Start (baseline) and end of intervention (week 8).
  Exploratory investigation of the Maternal Foetal Attachment Scale. The Maternal Foetal Attachment Scale has 24 items. The items are scored on a five-point scale (1-5) with a total score ranging from 24 to 120, with higher scores indicating greater maternal-foetal attachment.
To assess the effectiveness of group prenatal yoga to increase mother-foetal attachment | Start (baseline) and end of intervention (week 8).
  Exploratory investigation of the Maternal Antenatal Attachment Scale. The Maternal Antenatal Attachment Scale has a scale range of 1-5 with a total score ranging from 19-95, with higher scores indicating greater maternal antenatal attachment.
To assess whether yoga improves further aspects of mental health | Start (baseline) and end of intervention (week 8).
  The Edinburgh Postnatal Depression Scale (EPDS). The Edinburgh Postnatal Depression Scale (EPDS) has a range of 0-3, with a scale total range of 0-30, where higher scores indicate greater depressive symptoms.
To assess whether yoga improves further aspects of mental health | Start (baseline) and end of intervention (week 8).
  Beck Depression Inventory (BDI). The Beck Depression Inventory (BDI) has a scale range of 0-63, with higher scores indicating greater depressive symptoms. Each answer is scored on a scale value of 0-3.
To assess whether yoga improves further aspects of mental health | Start (baseline) and end of intervention (week 8).
  State and Train Anxiety Inventory (STAI). The State and Trait Anxiety Inventory (STAI) is rated on a 4-point Likert scale and has a total scale range of 20-80, with higher scores indicating greater anxiety symptoms.
To assess whether yoga improves further aspects of mental health | Start (baseline) and end of intervention (week 8).
  Perceived Stress Scale (PSS). The PSS questionnaire typically contains 10 questions, and respondents rate their feelings and thoughts over the past month on a 5-point scale. The Perceived Stress Scale (PSS) has a scale range of 0-40, where higher scores indicate greater perceived stress.
To ascertain whether yoga affects mother-infant bond (postpartum) | Start (baseline) and end of intervention (week 8).
  Maternal Attachment Inventory (MAI). The Maternal Attachment Inventory (MAI) has a scale range of 22-88, with higher scores indicating greater maternal attachment.
To ascertain whether yoga improves social support and efficacy | Start (baseline) and end of intervention (week 8).
  Multidimensional Scale of Perceived Social Support (MSPSS). The Multidimensional Scale of Perceived Social Support (MSPSS) has a total scale range of 12-84 or subscale ranges of 3-7, with higher scores indicating greater perceived social support.
To ascertain whether yoga improves social support and efficacy | Start (baseline) and end of intervention (week 8).
  The Short General Self-Efficacy Scale (GSE-6). The Short General Self-Efficacy Scale (GSE-6) has a scale range of 6-30, with higher scores indicating greater general self-efficacy.
To identify how the yoga sessions affect the lived experience of ethnic minority pregnant women | End of intervention (week 8).
  Focus groups
To identify how the yoga sessions are perceived by the yoga teachers | End of intervention (week 8).
  Interviews
To assess the effectiveness of group prenatal yoga to increase mother-foetal attachment | Start (baseline) and end of intervention (week 8).
  Changes in scores of the Prenatal Attachment Inventory. The Prenatal Attachment Inventory has 21 items and is a scale ranging from 21-84, with higher scores indicating greater prenatal attachment.
  items

CONTACTS AND LOCATIONS:
Locations (1):
- Maurice Wohl Clinical Neuroscience Institute, 5 Cutcombe Rd, Brixton, London SE5 9RT, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Estevao C, Chiarpenello C, Kwok W, Bhargav H, Jasti N, Chandra P, Varambally S, Pariante C. Co-designing and evaluating a prenatal yoga intervention for ethnic minority women: a feasibility study. Pilot Feasibility Stud. 2025 Jul 7;11(1):96. doi: 10.1186/s40814-025-01667-9. PMID 40624724